CLINICAL TRIAL: NCT06275633
Title: Behavioural Profiling of Disease-related Cognitive and Motor Impairment With Focus on Dopaminergic Effects in Parkinson's Disease and Potential Correlation to Biomarkers.
Brief Title: Behavioural Profiling of Disease-related Cognitive and Motor Impairment in PD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Bispebjerg and Frederiksberg (Other)
Responsible Party: Principal Investigator, Annemette Lokkegaard, Associate professor, University Hospital Bispebjerg and Frederiksberg
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: H-18055648
Record Dates: First submitted 2023-09-14; First posted 2024-02-23 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Parkinson Disease; Medication; UPDRS; Motor Function; Cognitive Impairment; Depression; Impulsive; Levodopa
MeSH Terms: conditions — Parkinson Disease; Cognitive Dysfunction; Depression; Impulsive Behavior | interventions — Levodopa

STUDY DESIGN:
Intervention Model Description: This is a prospective patient with Parkinson's Disease cohort. After acute levodopa challenge test patients with Parkinson's Disease are divided due to measured levodopa response and their self-rated medicine effect.
Masking Description: There will be a blinded assessment of videos of participants with Parkinson's Disease ON and OFF medication
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Effect of levodopa (Experimental): 1. Patients with PD are first being tested "off medication"
  2. After examination OFF, the same group is being tested after adm of 200 mg Madopar Q
  Interventions: Drug: Levodopa

INTERVENTIONS:
Drug: Levodopa — Medicine response

SUMMARY:
In this project, patients with Parkinson's Disease (PD) will be characterized by measuring cognitive and motor function and relation to effect of Levodopa.

Participants will be patients with Parkinson's Disease and healthy controls. It will be investigated if there is a difference between patients with a good measured Levodopa response and with a poor measured response.

DETAILED DESCRIPTION:
The patients with Parkinson's Disease will be included from the outpatient clinic at the Department of Neurology at Bispebjerg Frederiksberg Hospital and healthy controls will be found among relatives or volunteers through research ads.

Patients will be asked to pause dopaminergic medication for 6 half times.Then a baseline examination will be performed in the morning in a non-medicated state (OFF), using Unified Parkinson's disease rating Scale (UPDRS), the MOntreal Cognitive Assessment (MoCA) and computerized cognitive testing. Baseline screening for depression with Beck Depression Inventory (BDI) and for impulsivity with Questionnaire for Impulsive-Compulsive Disorders in Parkinson's Disease-Rating Scale (QUIP).

An acute levodopa challenge will be performed with patients receiving 200/25 mg dispersible levodopa/benserazide. After an hour UPDRS and cognitive computerized tests are repeated.

This is estimated to take about 3½ hours to complete. In healthy controls a neurological examination, BDI and MoCA will pe performed.

The UPDRS motor test is videotaped. A specialist will later evaluate the motor function blinded.

The participants will be asked to participate in the Bispebjerg Frederiksberg (BFH) BioBank, BFH-2017-114, (ISuite nr.: 05991) at Bispebjerg Frederiksberg Hospital for future research.

An exact calculation of power is difficult to calculate as the project includes a broad range of correlations.

Numeric data will be analysed using the Student's t-test (when normal distribution is met) or Wilcoxon rank sum test (when normal distribution is not met). Binary data will be analysed using the Fishers exact test.

ELIGIBILITY:
Inclusion Criteria:

* Age of minimum 18
* Diagnosis of PD
* Be able to cooperate, understand and participate in the project
* Signed informed consent, including consent to being included in the Biobank

Exclusion Criteria:

* Dementia
* Treatment with anti-dopaminergic medication.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — "Sex" means a person's classification as male or female based on biological distinctions.
Enrollment: 68 (Actual)
Dates: Start 2019-03-19 (Actual); Primary Completion 2021-12-03 (Actual); Study Completion 2023-07-30 (Actual)

PRIMARY OUTCOMES:
Motor improvement | Baseline to end of Levodopa challenge test, approximately 3-4 hours
  Unified Parkinson's disease rating scale, motor part (UPDRS-3) OFF medication compared to ON medication

SECONDARY OUTCOMES:
Cognitive function | Baseline to end of Levodopa challenge test, approximately 3-4 hours
  Cognitive computer tests

OTHER OUTCOMES:
Cognitive function | Baseline
  The Montreal Cognitive Assessment (MoCA)
Depressive symptoms | Baseline
  BDI, Beck Depression Inventory
Impulsivity | Baseline
  QUIP, Questionnaire for Impulsive-Compulsive Disorders in Parkinson's Disease-Rating Scale

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Bispebjerg and Frederiksberg, Copenhagen, Capital Region, Denmark